CLINICAL TRIAL: NCT03849456
Title: Safety and Tolerability of GWP42006 in Children and Young Adults With Autism Spectrum Disorder
Brief Title: Safety and Tolerability of Cannabidivarin (CBDV) in Children and Young Adults With Autism Spectrum Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to enrollment challenges during COVID-19 pandemic.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWND18089
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Cannabidivarin; CBDV; GWP42006
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — cannabidivarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GWP42006 (Experimental): Oral solution taken twice daily with food for 52 weeks.
  Interventions: Drug: GWP42006

INTERVENTIONS:
Drug: GWP42006 — Oral solution containing cannabidivarin 50 milligrams per milliliter (mg/mL) in sesame oil with anhydrous ethanol, sucralose, strawberry flavoring, and β-carotene.
  Other Names: Cannabidivarin; CBDV

SUMMARY:
To determine the safety and tolerability of GWP42006 (cannabidivarin, CBDV) in children and young adults with autism spectrum disorder (ASD) and to examine the effect of GWP42006 on communication, social interactions, sleep, behavior, and cognition profiles.

DETAILED DESCRIPTION:
This is a 52-week, open-label trial to evaluate the safety and tolerability of GWP42006. Participants who satisfy all eligibility criteria will start GWP42006 at a dose of 2.5 milligrams per kilogram per day (mg/kg/day) and titrate to a target dose of 10 mg/kg/day or 800 mg/day, whichever is smaller, during the first 4 weeks of treatment. If there is intolerance during titration, the participant may be maintained on a dose below 10 mg/kg/day. The maximum dose participants aged 6 years or older can receive will be 20 mg/kg/day or 1600 mg/day, whichever is smaller. Following the final treatment dose, participants will taper GWP42006 10% per day. The investigator will withdraw participants who fail to demonstrate any perceived benefit and may withdraw participants for whom tolerability is poor.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder (ASD) as defined by the Autism Diagnostic Observation Schedule, 2nd Edition and The Diagnostic and Statistical Manual of Mental Disorders, 5th Edition
* Intelligence quotient (IQ) of 40-120 (inclusive)
* Participant and their caregiver are English speaking.
* In the opinion of the investigator, the participant presents with ASD symptoms that warrant a therapeutic trial with GWP42006.

Key Exclusion Criteria:

* Known single gene neurogenetic disorder with high rates of epilepsy/autism (e.g., fragile X, tuberous sclerosis complex), structural brain lesion (prior stroke or hemispheric brain malformations), or history of any other epileptic encephalopathy, including infantile spasms, before the diagnosis of ASD
* More than 2 epileptic seizures per month within the 6 months prior to screening
* Initiation of a behavioral therapy program, new psychotropic medication, or therapeutic diet within the 2 months prior to screening, or plan to change or start any of the above during the trial
* Presence of a significant untreated medical problem (obstructive sleep apnoea, restless legs syndrome, gastroesophageal reflux disease, etc.) which may have significant impact on sleep study measures
* Behavioral management issues (e.g., self-injury, aggression) severe enough to be of safety concerns (to participant and/or staff)
* Clinically significant electrocardiogram abnormality or postural drop in systolic blood pressure at screening
* Any known or suspected hypersensitivity to cannabinoids or any of the excipients of GWP42006, such as sesame oil
* Known history of psychiatric disorder (defined as schizophrenia, bipolar disorder, or other psychiatric disease with a known history of hallucinations or delusions)
* History of any inborn errors of metabolism
* Significantly impaired hepatic function at screening
* Received an investigational product within the 3 months prior to screening
* Participant has been taking felbamate for less than 1 year prior to screening
* History of substance use disorders or positive drug of abuse dipstick test at screening (unless the positive result is due to a known concomitant medication)
* Currently using or has used recreational or medicinal cannabis or cannabinoid-based medications within the 3 months prior to screening and is unwilling to abstain for the duration of the trial
* Any history of suicidal behavior or any suicidal ideation within the month prior to or at screening

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experienced Severe Treatment-Emergent Adverse Events (TEAEs) | Day 1 to Day 403
  A TEAE was defined as an adverse event (AE) with an onset date on or after the first dose of GWP42006. If an AE had a partial onset date and it was unclear from the partial date (or the stop date) whether the AE started prior to or following the first dose of GWP42006, then the AE was considered a TEAE. The number of participants who experienced one or more severe TEAEs after dosing on Day 1 through to the Safety Follow-up will be presented.

SECONDARY OUTCOMES:
Change from Baseline in Children's Communication Checklist-2 (CCC-2) | Baseline to End of Treatment (Day 365) or Early Termination (ET)
  The CCC-2 is a caregiver-completed measure designed to assess the communication skills of children 4 to 16 years of age. An increase in score indicates an improvement.
Change from Baseline in Social Responsiveness Scale-2 (SRS-2) | Baseline to End of Treatment (Day 365) or ET
  The SRS-2 assesses social impairment associated with Autism Spectrum Disorder (ASD). Total scores between 58 and 72 indicate a mild deficiency, between 73 and 97 indicate a moderate deficiency, and 98 or above indicate a severe deficiency. A decrease in total score indicates an improvement.
Change from Baseline in Vineland Adaptive Behavior Scales, 3rd Edition (Vineland-3) | Baseline to End of Treatment (Day 365) or ET
  The Vineland-3 measures the personal and social skills of individuals from birth through adulthood. Score ranges are as follows: 70 to 80, borderline adaptive functioning; 51 to 70, mildly deficient adaptive functioning; 35 to 50, moderately deficient adaptive behavior; 20 to 35, severely deficient adaptive behavior; less than 20, markedly or profoundly deficient adaptive behavior.
Change from Baseline in National Institutes of Health (NIH) Toolbox Cognition Battery | Baseline to End of Treatment (Day 365) or ET
  The NIH Toolbox Cognition Battery has computerized instruments that measure several ability subdomains important for cognitive health.
Change from Baseline in Repetitive Behavioral Scale - Revised (RBS-R) | Baseline to End of Treatment (Day 365) or ET
  The RBS-R is used to measure the breadth of repetitive behavior in children, adolescents, and adults with ASD. Total scores range from 0 to 129. A decrease in total score indicates an improvement.
Change from Baseline in Children's Sleep Habits Questionnaire (CSHQ) | Baseline to End of Treatment (Day 365) or ET
  The CSHQ is used to examine sleep behavior in young children. Responses are given on a 5-point scale (1 = always; 5 = never). A higher score reflects more sleep problems.
Change from Baseline in Aberrant Behavior Checklist (ABC) | Baseline to End of Treatment (Day 365) or ET
  The ABC assesses the presence and severity of various problem behaviors commonly observed in individuals diagnosed with intellectual and developmental disabilities. Total scores range from 0 to 174. A decrease in total score indicates an improvement.
Clinical Global Impressions-Improvement (CGI-Improvement) | Baseline to End of Treatment (Day 365) or ET
  The CGI-Improvement evaluates the change from the initiation of treatment in the severity of psychopathology using a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Lower scores represent an improvement.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clinical Trial Site, Louisville, Kentucky
  - Clinical Trial Site, Lexington, Massachusetts
  - Clinical Trial Site, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No